CLINICAL TRIAL: NCT00263744
Title: A Phase I/II Study to Evaluate the Safety and Immunogenicity of MEDI-517, a Virus-Like Particle Vaccine Against Human Papillomavirus (HPV) Types 16 and 18, in Healthy Adult Female Volunteers Who Are HPV-16 or HPV-18 DNA Positive
Brief Title: Study to Evaluate the Safety and Immunogenicity of MEDI-517P in Healthy Adult Female Volunteers Who Are HPV-16 or HPV-18 DNA Positive
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Genevieve Lonosky, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MI-CP058
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
MeSH Terms: interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MEDI517
  Interventions: Biological: MEDI 517
- 2 (Active Comparator): Aluminum hydroxide
  Interventions: Other: Aluminum hydroxide

INTERVENTIONS:
Biological: MEDI 517 — Vaccine is supplied in single use vials containing 0.75 mL of MEDI-517 at a concentration of 40 mg/0.5 mL formulated with SBAS4 adjuvant.
  Arms: 1
Other: Aluminum hydroxide — Aluminum hydroxide supplied in single use vials containing 0.75 mL of aluminum hydroxide at a concentration of 0.5 mg of aluminum in the form of aluminum hydroxide per 0.5 mL.
  Arms: 2

SUMMARY:
The primary objective of this study is to describe the safety of 40 mg MEDI-517, with a control of aluminum hydroxide, when given to healthy adult women who have evidence of HPV-16 and/or HPV-18 DNA detected in cervical brushings.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 through 30 years of age (must not have reached the 31st birthday)
* Unless previously surgically sterilized, agrees to use an effective method of birth control (e.g., abstinence, intrauterine contraceptive device, oral contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam, Norplant® or DepoProvera®) beginning 30 days before the first study injection and continuing through 60 days after the final study injection
* Healthy by medical history and physical examination
* Cervical specimen positive for HPV-16 and/or HPV-18 DNA using the Digene Hybrid Capture® II HPV test within 21 days of study entry
* Cervical cytology by Pap smear that is either normal or no greater than ASCUS or AGCUS, using the Cytyc ThinPrep® Pap Test, within 21 days of study entry (a normal Pap smear must also be adequate for interpretation; a Pap smear that is normal but inadequate for interpretation must be repeated). Those volunteers with ASCUS or AGCUS must have had a clinical evaluation by colposcopy within the previous month which showed no evidence of CIN or SIL.
* No evidence of anogenital HPV lesions or no physical findings suggestive of other gynecologic pathogens on pelvic examination within 21 days of study entry
* Agrees to no other experimental therapy or vaccines until 30 days after the last study injection
* Written informed consent obtained from the volunteer

Exclusion Criteria:

* Acute illness or fever (oral temperature ³99.5°F [37.5°C]) at start of the study
* History or clinical manifestations of significant medical or psychiatric disorder
* Pregnant or lactating
* Use of immunosuppressive medication (inhaled and topical corticosteroids are permitted) within the previous 90 days or history of immunodeficiency
* History of cancer
* History of alcohol or drug abuse within the past 2 years
* At screening (must be within 21 days of study entry) any of the following: hemoglobin <11 gm/dL; white blood cell count <4000/mm3; platelet count <120,000/mm3; AST, ALT, creatinine >1.5x upper limit of normal for the laboratory in question; other abnormal laboratory values in the screening panel which in the opinion of the principal investigator are judged to be clinically significant
* Receipt of immunoglobulin or blood products within 90 days prior to study entry
* History of Pap smear more severe than ASCUS or AGCUS
* Positive tests for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 antibody
* Any prior receipt of any vaccine or therapy (experimental or otherwise) for treatment or prophylaxis of genital warts or other papillomavirus related condition. Any treatment of genital warts or other papillomavirus related condition within six months of randomization (local therapy for common skin and/or plantar warts is allowed)
* Prior receipt of any vaccine containing monophosphoryl lipid A or SBAS4 adjuvant (no vaccines currently licensed contain these)
* Receipt of any experimental vaccine within 90 days prior to entry into this study
* Receipt of any experimental drug therapy within 30 days or five half-lives of the experimental drug (if the half-life is known), whichever is longer

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 1999-11; Primary Completion 2001-04 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety in terms of unsolicited adverse events and serious adverse events. | 7 days after each injection

SECONDARY OUTCOMES:
Determine the effect of MEDI-517 compared to aluminum hydroxide control on the proportion of volunteers who are positive for HPV DNA. | Swab taken on Study Day 210

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Losonsky, M.D., Study Director — MedImmune LLC